CLINICAL TRIAL: NCT05984992
Title: A Randomized, Double-blinded, Placebo-controlled, Single Ascending Dose Study to Assess the Safety, Tolerability and Pharmacokinetics of SRN-001 in Healthy Participants
Brief Title: The First-in-human Study of SRN-001 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: siRNAgen Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SRN-001-C01
Record Dates: First submitted 2023-07-26; First posted 2023-08-09 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-10

CONDITIONS: Idiopathic Pulmonary Fibrosis
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis

STUDY DESIGN:
Intervention Model Description: Randomized, Double-blinded, Placebo-controlled, Single Ascending Dose
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SRN-001 (Experimental)
  Interventions: Drug: SRN-001
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SRN-001 — siRNA therapeutics, Self Assembled Micelle inhibitory RNA platform utilized
  Arms: SRN-001
Drug: Placebo — 0.9% Sodium Chloride(Normal saline)
  Arms: Placebo

SUMMARY:
SRN-001 is a novel small interfering RNA (siRNA) drug being developed to treat fibrosis using Self Assembled Micelle inhibitory ribonucleic acid (SAMiRNA™) technology. Amphiregulin (AREG) is a growth factor involved in fibroblast proliferation and myofibroblast transformation which is the hallmark of fibrosis in lung and kidney tissues. AREG is a downstream gene overexpressed by Transforming growth factor-β (TGF-β) during fibrosis, promoting fibroblast to myofibroblast transition (FMT). SRN-001 is designed to downregulate generating amphiregulin by RNA interference (RNAi). The goal of this clinical trial is to evaluate safety, tolerability, and pharmacokinetics in healthy participants. This trial is first-in-human clinical trial to develop SAMiRNA™ to utilize as therapeutic use.

DETAILED DESCRIPTION:
Participants with part in consent will be enrolled in a phase 1a study of SRN-001. Prior to initiation of treatment, participants will undergo several screening test for checking their condition of health. There is no specific test comparing with the general other clinical trial in healthy volunteers. They will be randomized into two groups, active drug and inactive placebo(normal saline) as ratio 2:1. Starting dose is planned 15mg. For confirming maximal tolerable dose, dose will be escalated when no dose-limiting toxicity (DLT) confirmed. Each cohort will take single dose and for 4 weeks, safety observation will be taken. If safety abnormality will be retained in 4 weeks, the participant's safety observation will be prolonged by the end of the adverse event once 2 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-70
* BMI ≥18.0 kg/㎡ and ≤35 kg/㎡
* 12-lead triplicate electrocardiogram (ECG) readings within normal limits or with no clinically significant abnormalities
* systolic blood pressure ≥ 90 mmHg and ≤160 mmHg; a diastolic blood pressure ≥ 50 mmHg and ≤95 mmHg; pulse ≥ 45 bpm and ≤100 bpm; tympanic temperature ≥ 35.5°C and ≤37.7°C and respiratory rate 12rpm to 22rpm
* Negative urinary cotinine
* Compliance to contraception and sperm donation restriction
* Participants who are able and willing to give written informed consent
* Fully vaccinated against SARS-CoV-2

Exclusion Criteria:

* Who has clinically significant history
* Who is with history of multiple drug allergies or history of allergic reaction to an oligonucleotide or common medicine (eg, aspirin, antibiotics, etc) or clinically significant hypersensitivity
* No tolerance to IV injections or significant potential of intolerance
* Clinically significant surgical history within 1 year
* History of drug abuse or alcoholism within 2 years, and a restriction of consuming alcohol during study period
* Pregnant or lactating females
* Liver function test is 1.5 times greater than upper limit of normal (ULN)
* Albumin ≥ 35 g/L and ≤ 50 g/L
* Hb < 115 g/L (female), < 125 g/L (male)
* estimated glomerular filtration rate (eGFR) < 60 mL/min (CKD-EPI), 90 mL/min (MDRD)
* Glucose < 3 mmol/L
* Positive screen for alcohol or drugs of abuse
* HBsAg, Hepatitis B virus (HBV), Hepatitis C virus (HCV), or HIV infection
* QTcF > 450 msec for male, > 470 msec for female
* Inappropriate lab result by physician's discretion
* Who have donated > 500 mL of blood within 3 months
* Who have received an investigational agent within 3 months, or 5 half-lives
* Who have used prescription medication within 4 weeks including vaccines
* Who have used OTC medication within 7 days
* With clinically relevant wounds, following a clinically relevant surgery or have recently completed any invasive procedures (ie, Endoscopy) within 1 week, or who are scheduled for an elective surgical procedure
* Who have a significant infection or known inflammatory process ongoing
* Any conditions that, in physician's opinion, would make the participant unsuitable for enrollment or could interfere with the participant's participation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2023-09-08 (Actual); Primary Completion 2024-03-15 (Actual); Study Completion 2024-09-25 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-emergent adverse events(TEAEs) | Up to 4 weeks
Number of participants with serious adverse events(SAEs) | Up to 4 weeks

SECONDARY OUTCOMES:
Cmax | Up to 168 hours post-dose
  Maximum observed concentration
Clast | Up to 168 hours post-dose
  Observed concentration corresponding to Tlast
Tlast | Up to 168 hours post-dose
  Time of last measurable observed concentration
AUClast | Up to 168 hours post-dose
  Area under the drug concentration-time curve, from time zero to the last measurable concentration
AUCinf | Up to 168 hours post-dose
  Area under the drug concentration-time curve, from time zero to infinity
T½ | Up to 168 hours post-dose
  Apparent terminal half-life
Kel | Up to 168 hours post-dose
  Apparent terminal elimination rate constant
CL | Up to 168 hours post-dose
  Total body clearance
Vz | Up to 168 hours post-dose
  Volume of distribution
MRT | Up to 168 hours post-dose
  Mean residence time

OTHER OUTCOMES:
Incidence of treatment-emergent Anti-Drug Antibody(ADA) | Up to 672 hours post-dose
Change from baseline in specific biomarkers | Up to 24 hours post-dose

CONTACTS AND LOCATIONS:
Locations (1):
- CMAX Clinical Research, Adelaide, South Australia, Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gleason DF, Mellinger GT. Prediction of prognosis for prostatic adenocarcinoma by combined histological grading and clinical staging. J Urol. 1974 Jan;111(1):58-64. doi: 10.1016/s0022-5347(17)59889-4. No abstract available. PMID 4813554
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/26817844/